CLINICAL TRIAL: NCT02562313
Title: A Trial Investigating the Continuous Subcutaneous Insulin Infusion of a Liquid Formulation of BioChaperone Insulin Lispro in Comparison to Humalog®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BC3-CT015
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BioChaperone insulin lispro (Experimental)
  Interventions: Drug: BioChaperone insulin lispro
- Humalog® (Active Comparator): Insulin lispro
  Interventions: Drug: Humalog®

INTERVENTIONS:
Drug: BioChaperone insulin lispro — BioChaperone insulin lispro bolus infusion followed by test meal intake
  Arms: BioChaperone insulin lispro
Drug: Humalog® — Humalog® bolus infusion followed by test meal intake
  Arms: Humalog®

SUMMARY:
This study is constituted of 2 parts:

Part A: A total of 36 patients will be enrolled in part A. Each eligible subject will participate in two 14-day treatment periods with Continuous Subcutaneous Insulin Infusion (CSII) of BioChaperone insulin lispro and insulin lispro (Humalog®, Eli Lilly and Company). Each treatment period consists of 10 treatment days under free living conditions (e.g. home / workplace) and under standardised conditions at the clinic. Various assessments for pharmacodynamics, pharmacokinetics, pump compatibility, short-term efficacy and safety are performed on selected days, including:

* Mixed Meal Test (MMT), Day 1, Day 3, Day 12 and Day 14, that will assess the post-prandial glucose response for 6 hours after individualized standard meal (fixed nutrient ratio) ingestion and bolus administration via CSII.
* Continuous Glucose Monitoring (CGM), (Day 1 - 14) that will be used in blinded mode (i.e. neither subjects nor the investigators are aware of the sensor glucose values).
* Pump compatibility (Day 1 - 14): Subjects will continue CSII treatment with the Investigational Medicinal Products (IMP) during the outpatient periods.

Part B: A total of 44 patients will be enrolled. Subjects will be randomized to a 4-period cross-over study aiming at comparing the performance of BC Lispro and Humalog after a prandial bolus administration with two different CSII systems (Roche Accu-Chek® Spirit and Medtronic Paradigm® Veo™) or with a syringe. Pharmacodynamics, pharmacokinetics, pump compatibility and safety will be analyzed.

Each period will include a mixed meal tolerance test with a CSII device and a mixed meal tolerance test with the same dose of insulin administered with a syringe.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Body Mass Index (BMI) between 18.5 and 28.5 kg/m^2, both inclusive
* Using or having used a Roche CSII system (Accu-Chek® Spirit Combo/ Accu- Chek® Spirit) for at least 6 months before screening. In Part B subjects using any form of CSII treatment for at least 6 months before screening will be included.
* HbA1c <= 9.0%.
* Total insulin dose of < 1.2 (I)U/kg/day
* Ability to calculate insulin bolus manually or using a bolus calculator and willingness to consume regular meals, perform carbohydrate counting, self-monitoring of plasma glucose (SMPG) profiles and use of Continuous Glucose Monitoring (CGM).
* Fasting C-peptide <= 0.30 nmol/L

Exclusion Criteria:

* Known or suspected hypersensitivity to Investigational Medicinal Product(s) (IMP(s)) or related products
* Type 2 diabetes mellitus
* Previous participation in this trial.
* Receipt of any investigational product in a clinical trial within 60 days before randomisation in this trial
* Clinically significant abnormal haematology, biochemistry, urinalysis, or coagulation screening test
* Presence of clinically significant acute gastrointestinal symptoms
* Known slowing of gastric emptying and or gastrointestinal surgery
* Unusual meal habits and special dietary requirements or unwillingness to eat the food provided in the trial
* History of diabetic ketoacidosis (DKA) episodes requiring hospitalization within 6 months prior to screening
* History of abscess at the infusion site within 6 months prior to screening
* Hypoglycaemia unawareness as judged by the Investigator
* History of severe hypoglycaemic episodes requiring hospitalization within the last 6 months prior to screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: ΔAUCBG 0-2h | 2 Hours
  Incremental Area Under the Blood Glucose concentration-time Curve from 0-2 hours after the start of the meal.
Pharmacokinetics: AUClis 0-30min | 30 minutes
  Area Under the serum insulin Lispro concentration-time Curve from 0-30 minutes

SECONDARY OUTCOMES:
AUClis_0-6h | up to 6 Hours
  Area Under the baseline adjusted insulin Lispro Curve from 0-6h following a bolus dose
Cmax | up to 6 Hours
  Maximum insulin Concentration following a bolus dose
tCmax | up to 6 Hours
  Time to Maximum insulin Concentration following a bolus dose
BGmax | up to 6 Hours
  Maximum Blood Glucose after start of an individualised standardised meal intake
tBGmax | up to 6 Hours
  Time to Maximum Blood Glucose concentration
Compatibility | up to 14 days
  Number of suspected episodes of infusion set occlusion or leakage
Adverse Events | up to 12 weeks
  Number of Adverse Events
Local tolerability | up to 12 weeks
  Number of injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil GmbH
Locations (1):
- Profil GmbH, Neuss, Germany